CLINICAL TRIAL: NCT00890799
Title: Clinical Evaluation of Transcatheter Closure and Surgery of Perimembranous Ventricular Septal Defects
Brief Title: Transcatheter Closure Versus Surgery of Perimembranous Ventricular Septal Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Jian Yang, Dr Jian Yang, Xijing Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: XJ-20090315
Record Dates: First submitted 2009-04-23; First posted 2009-04-30 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Ventricular Septal Defects
Keywords: transcatheter closure; ventricular septal defects
MeSH Terms: conditions — Heart Septal Defects, Ventricular | interventions — Surgical Procedures, Operative; Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- occluders (Experimental): Shanghai pmVSD occluder (LEPU Medical Tech-nology Co, Ltd, Beijing, China) was used in this study.
  Interventions: Device: Shanghai pmVSD occluder; Procedure: surgery

INTERVENTIONS:
Device: Shanghai pmVSD occluder — Ventricular Septal Defects Occluders with sizes from 4mm to 20mm.
  Other Names: Shanghai pmVSD-O
Procedure: surgery — Patient in this group received open surgical repair of pmVSD.
  Other Names: open surgery

SUMMARY:
The purpose of this study is to investigate effectiveness and safety of transcatheter closure of perimembranous ventricular septal defects.

DETAILED DESCRIPTION:
Perimembranous Ventricular septal defect (VSD) is the most common congenital cardiac malformation and constitutes over 20% of all congenital cardiac disease. Though conventional surgery for VSD is a widely accepted procedure with minimal operative mortality, it carries a small but definite risk of morbidity and mortality associated with cardiopulmonary bypass and surgical closure. The newly appeared transcatheter device closure technique provides an alternative to surgical closure. However, the mid-to-long term effects of this technique using occluders is not clear. The aim of this study was to evaluate the safety and effectiveness of transcatheter closure of perimembranous ventricular septal defects using septal occluders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ventricular septal defects eligible for transcatheter closure.

Exclusion Criteria:

* Patients less than 2 years old. Patients not suitable for transcatheter closure. Patients comorbid with other diseases.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Major adverse events | till study end
  Major adverse events included but were not limited to death during or after the procedure because of complications of the procedure,cAVB requiring pacemaker implantation, thromboembolism, and new-onset valvular regurgitation requiring surgical repair.

SECONDARY OUTCOMES:
Minor adverse events | Till study end
  Minor adverse events included but were not limited to groin hematoma, blood loss requiring transfusion, device embolization with transcatheter removal, any cardiac arrhythmia that required medication, new or increased valvular regurgitation less than two grades, hemolysis requiring medication, fever >38.5°C, rash, and loss of peripheral pulse. These minor adverse events required medical intervention but were not life threatening; they had no long-term sequelae and did not require long-term therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yang, M.D., Ph. D., Principal Investigator — Xijing Cardiovascular Hospital

REFERENCES:
- [Derived] Wang J, Zuo J, Yu S, Yi D, Yang X, Zhu X, Li J, Yang L, Xiong L, Ge S, Ren J, Yang J. Effectiveness and Safety of Transcatheter Closure of Perimembranous Ventricular Septal Defects in Adults. Am J Cardiol. 2016 Mar 15;117(6):980-7. doi: 10.1016/j.amjcard.2015.12.036. Epub 2015 Dec 31. PMID 26796197
- [Derived] Yang J, Yang L, Yu S, Liu J, Zuo J, Chen W, Duan W, Zheng Q, Xu X, Li J, Zhang J, Xu J, Sun L, Yang X, Xiong L, Yi D, Wang L, Liu Q, Ge S, Ren J. Transcatheter versus surgical closure of perimembranous ventricular septal defects in children: a randomized controlled trial. J Am Coll Cardiol. 2014 Apr 1;63(12):1159-1168. doi: 10.1016/j.jacc.2014.01.008. Epub 2014 Feb 5. PMID 24509270
- [Derived] Yang J, Yang L, Wan Y, Zuo J, Zhang J, Chen W, Li J, Sun L, Yu S, Liu J, Chen T, Duan W, Xiong L, Yi D. Transcatheter device closure of perimembranous ventricular septal defects: mid-term outcomes. Eur Heart J. 2010 Sep;31(18):2238-45. doi: 10.1093/eurheartj/ehq240. Epub 2010 Aug 27. PMID 20801925